CLINICAL TRIAL: NCT00435994
Title: Assessment of Airway Obstruction in Infants With Lower Respiratory Infections
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University School of Medicine (Other)
Collaborators: Thrasher Research Fund (Other)
Responsible Party: Sponsor
Organization: Indiana University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0311-21
Record Dates: First submitted 2007-01-25; First posted 2007-02-16 (Estimated); Results first posted 2016-06-01 (Estimated); Last update posted 2016-06-01 (Estimated); Status verified 2016-05

CONDITIONS: Bronchiolitis; Respiratory Syncytial Virus Infections
Keywords: Infant; Respiratory Syncytial Virus; Bronchiolitis
MeSH Terms: conditions — Bronchiolitis; Respiratory Syncytial Virus Infections | interventions — Epinephrine; Nasal Lavage Fluid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Infants with viral lower respiratory infections (Other): Infants between the ages of 2-24 month, with viral lower respiratory infection defined as first episode of wheezing and shortness of breath preceded by an upper respiratory tract infection, including hospitalized infants
  Interventions: Drug: Inhaled primatene will be given as a breathing treatment; Other: Nasal Washing
- Healthy Control (Other): Healthy infants between the ages of 2-24 month
  Interventions: Drug: Inhaled primatene will be given as a breathing treatment; Other: Nasal Washing
- Bronchiolitis-Nasal wash only (Other): Infants 2 months to 24 months who were diagnosed with bronchiolitis received nasal wash only
  Interventions: Other: Nasal Washing

INTERVENTIONS:
Drug: Inhaled primatene will be given as a breathing treatment — While the research subject is sedated an inhaled mist of primatene mist will be given to the patient.
  Other Names: epinephrine 0.5ml of the 2.25% concentration
  Arms: Healthy Control; Infants with viral lower respiratory infections
Other: Nasal Washing — 1-3 mls of normal saline will be instilled into the infant's nose and then aspirated to obtain the nasal fluid, which will be analyzed for VEGF level by ELISA and viral antigens by immunoflourescence

SUMMARY:
The purpose of this study is to evaluate how two different aerosol medications may improve airway function in infants with respiratory illness. We are using two different medications and comparing the difference in lung function after each medication. We will also be taking a nasal wash sample for VEGF. We will be using this in comparing how infants respond to the aerosol medications as well. We hope to help standardize medications used for infants with bronchiolitis and RSV.

DETAILED DESCRIPTION:
We hypothesize that VEGF production is higher in children with RSV infection than in children with other viral infections and normal controls. In addition, the degree of VEGF production is related to severity of airway obstruction. We also hypothesize that infants with higher VEGF levels are more likely to improve lung function following racemic epinephrine than albuterol.

ELIGIBILITY:
Inclusion Criteria:

* Group 1 Infants between 2 and 24 months that are healthy
* Group 2 Infants between 2 and 24 months that have RSV or bronchiolitis and defined as the first episode of wheezing

Exclusion Criteria:

* Group 1 and 2 - no cardiac disease, no oxygen requirement, prematurity < 37 weeks, and cannot be in the ICU.

Ages: 2 Months to 2 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 59 (Actual)
Dates: Start 2003-12; Primary Completion 2009-03 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert S. Tepper, MD, Principal Investigator — Indiana University
Locations (1):
- Riley Hospital for Children, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Control: Healthy infants between the ages of 2-24 month without a history of congenital heart disease or prematurity
- Respiratory Syncytial Virus: Infants between the ages of 2-24 month, with viral lower respiratory infection defined as first episode of wheezing and shortness of breath preceded by a URI
Period: Overall Study
Arm/Group | Healthy Control | Respiratory Syncytial Virus | Bronchiolitis-Nasal Wash Only
Started | 22 | 25 | 12
Completed | 15 (7 of the subjects were consented and did not complete the study procedures.) | 25 | 12
Not Completed | 7 | 0 | 0
Not completed — Lost to Follow-up | 7 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Bronchiolitis: Infants 2 months to 24 months who were diagnosed with bronchiolitis received nasal wash only.
- Total: Total of all reporting groups
Arm/Group | Healthy Control | Respiratory Syncytial Virus | Bronchiolitis | Total
Number analyzed (Participants) | 22 | 25 | 12 | 59
Age, Continuous [Mean (Standard Deviation); unit: months] | 13 (5) | 7 (6) | 7 (4) | 11 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 4 | 20
  Male | 13 | 18 | 8 | 39
Region of Enrollment [Number; unit: participants]
  United States | 22 | 25 | 12 | 59

OUTCOME MEASURES:

1. Primary Outcome: Lung Function
Description: Lung functions were obtained under sedation using Chloral Hydrate. Forced expiratory flows are a lung volume at which the airway pressure is equal to 30 cm H2O (V30). Forced expiratory flows are measured at 75% FVC (FEF75). Measurements were repeated post bronchodilator and again post Epinephrine. A higher Z-score reflects better lung function.
Time Frame: Baseline, Post bronchodilator (up to 10 minutes, Post-epinephrine (up to 30 minutes)
Population: All participants who had baseline, post bronchodilator and post epinephrine measurements were included. Participants in the Bronchiolitis arm did not have infant pulmonary functions obtained.
Measure: Mean (Standard Deviation); unit: Z score
Groups:
- Healthy Control: Healthy infants between the ages of 2-24 month without a history of congenital heart disease or prematurity had spirometry performed under sedation.
Arm/Group | Healthy Control | Respiratory Syncytial Virus
Number analyzed (Participants) | 10 | 3
Z score
  Baseline | 0.071 (0.586) | -3.179 (2.610)
  Post Bronchodilator | 0.186 (0.639) | -3.345 (2.112)
  Post Epinephrine | 0.041 (0.802) | -2.430 (2.716)
Statistical Analysis 1: Comparison: Healthy Control vs Respiratory Syncytial Virus; Test type: Superiority or Other; p = 0.0020, ANOVA

2. Primary Outcome: Endothelial Growth Factor (VEGF)
Description: Analysis for VEGF level by ELISA
Time Frame: During nasal wash
Population: Due to limited samples and the length of time that has passed since they were obtained, we are unable to separate Bronchiolitis from RSV.
Measure: Mean (Standard Deviation); unit: pg/dl
Groups:
- Bronchiolitis and Respiratory Syncytial Virus-Nasal Wash Only: Infants 2 months to 24 months who were diagnosed with bronchiolitis and respiratory syncytial virus received nasal wash only.
Arm/Group | Healthy Control | Bronchiolitis and Respiratory Syncytial Virus-Nasal Wash Only
Number analyzed (Participants) | 19 | 9
pg/dl | 183.526 (223.268) | 568.867 (407.257)
Statistical Analysis 1: Comparison: Healthy Control vs Bronchiolitis and Respiratory Syncytial Virus-Nasal Wash Only; Test type: Superiority or Other; p = .0020, ANOVA

ADVERSE EVENTS:
Arm/Group | Healthy Control | Respiratory Syncytial Virus | Bronchiolitis
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/25 | 0/12
Other Adverse Events (participants affected / at risk) | 0/15 | 0/25 | 0/12

LIMITATIONS AND CAVEATS:
More than half of our infants woke up before completion of the protocol therefore limiting our analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No